CLINICAL TRIAL: NCT01878942
Title: Psychological, Physiological, Endocrine, and Pharmacokinetic Effects of LSD in a Controlled Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK 279/12
Record Dates: First submitted 2013-05-27; First posted 2013-06-17 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: LSD; Pharmacology; Pharmacokinetics; Pharmacodynamics; Mechanism of action; Psychedelic; Serotonin; Prepulse inhibition; LSD-induced neuroendocrine effects; Long-term psychological effects
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Placebo, LSD (Other): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two treatment conditions in the same subject.
  Interventions: Drug: Placebo; Drug: LSD

INTERVENTIONS:
Drug: Placebo — Capsules containing mannitol looking identical to LSD
  per os
Drug: LSD — 200µg per os, single dose
  Other Names: Lysergic acid diethylamide

SUMMARY:
The purpose of this study is to characterize the acute psychological, physiological, endocrine, and pharmacokinetic, as well as long-term psychological effects of LSD in humans.

DETAILED DESCRIPTION:
Lysergic acid diethylamide (LSD) is the prototype hallucinogen used recreationally worldwide. In the 50-70s, LSD was also used to study psychotic-like states in normals ("model psychosis") and in "psycholytic psychotherapy". Potential research and therapeutic uses of LSD are now re-recognized and may include its use in brain research, treatment of cluster headache, and aid in psychotherapy and in terminally ill patients. A better and contemporary understanding of the pharmacology of LSD is important in the light of its widespread recreational, and potential scientific and therapeutic uses. The study has no primary therapeutic intentions but aims for a solid account of the clinical pharmacological characteristics of the drug. To characterize the acute physiological, psychological, endocrine, and pharmacological response to the administration of a single dose of LSD in healthy subjects the investigators use a randomized double-blind placebo-controlled cross-over design with two experimental sessions. Subjects will participate in a placebo and a LSD session. Subjective and cardiovascular responses will be repeatedly assessed throughout the experiments and plasma samples are collected for pharmacokinetics and endocrine measurements.Additionally long-term psychological changes associated with the LSD experience are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years
2. Understanding of the German language
3. Understanding the procedures and the risks associated with the study
4. Participants must be willing to adhere to the protocol and sign the consent form
5. Participants must be willing to refrain from taking illicit psychoactive substances during the study
6. Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session, as well as during the study day.
7. Participants must be willing not to drive a traffic vehicle within 48 h following LSD administration.
8. Women of childbearing potential must have a negative pregnancy test at the beginning of the study and must agree to use an effective form of birth control. Pregnancy tests are repeated before each study session.

Exclusion Criteria:

1. Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>150/95 mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder.
2. Current or previous psychotic or major affective disorder
3. Psychotic or major affective disorder in first-degree relatives
4. Relevant prior illicit drug use (except tetrahydrocannabinol (THC)-containing products) more than 10 times or any time within the previous 2 months.
5. Pregnant or nursing women.
6. Participation in another clinical trial (currently or within the last 30 days)
7. Use of medications that may interfere with the effects of the study medications (any psychiatric medications)
8. Insufficient interpersonal relationship/rapport with study physician as judged by the study physician

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-06; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Subjective / psychological effects of LSD | 24 hours
  repeated assessment of subjective effects with validated questionnaires

SECONDARY OUTCOMES:
Physiological effects of LSD | 24 hours
  Effect on blood pressure, heart rate, body temperature, and pupillary function
Endocrine response of LSD | 24 hours
Pharmacokinetics of LSD | 24 hours
  Time course of plasma concentration, half-life, pharmacokinetic-pharmacodynamic relationship
Effect of LSD on prepulse inhibition | 3 hours
  Pre-Pulse inhibition of the acoustic startle reflex
Tolerability of LSD | 24 hours
  Assessment of adverse effects
Long-term psychological effects of LSD | 12 months
  Assessment of long-term psychological effects after 1 and 12 months
Genetic Polymorphisms | assessed once, at time of screening visit or at time of end of study visit
  Effects of genetic polymorphisms on the response to LSD
Effects on social cognition and empathy | 8 h
  assessment of cognitive and emotional empathy, as well as of prosocial behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Schmid Y, Liechti ME. Long-lasting subjective effects of LSD in normal subjects. Psychopharmacology (Berl). 2018 Feb;235(2):535-545. doi: 10.1007/s00213-017-4733-3. Epub 2017 Sep 16. PMID 28918441
- [Derived] Dolder PC, Schmid Y, Steuer AE, Kraemer T, Rentsch KM, Hammann F, Liechti ME. Pharmacokinetics and Pharmacodynamics of Lysergic Acid Diethylamide in Healthy Subjects. Clin Pharmacokinet. 2017 Oct;56(10):1219-1230. doi: 10.1007/s40262-017-0513-9. PMID 28197931
- [Derived] Liechti ME, Dolder PC, Schmid Y. Alterations of consciousness and mystical-type experiences after acute LSD in humans. Psychopharmacology (Berl). 2017 May;234(9-10):1499-1510. doi: 10.1007/s00213-016-4453-0. Epub 2016 Oct 7. PMID 27714429
- [Derived] Dolder PC, Schmid Y, Muller F, Borgwardt S, Liechti ME. LSD Acutely Impairs Fear Recognition and Enhances Emotional Empathy and Sociality. Neuropsychopharmacology. 2016 Oct;41(11):2638-46. doi: 10.1038/npp.2016.82. Epub 2016 Jun 1. PMID 27249781
- [Derived] Schmid Y, Enzler F, Gasser P, Grouzmann E, Preller KH, Vollenweider FX, Brenneisen R, Muller F, Borgwardt S, Liechti ME. Acute Effects of Lysergic Acid Diethylamide in Healthy Subjects. Biol Psychiatry. 2015 Oct 15;78(8):544-53. doi: 10.1016/j.biopsych.2014.11.015. Epub 2014 Nov 29. PMID 25575620